CLINICAL TRIAL: NCT07075211
Title: Effect of Mini-screw Assisted Rapid Palatal Expansion on Midpalatal Suture in Post-pubertal Patients: a CBCT Study
Acronym: EMARPEMSPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aseel AlNaimi, postgraduate orthodontic student, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0803024OR
Record Dates: First submitted 2025-06-15; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Constricted Maxillary Arch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- participants who received MARPE (Experimental): participants who received MARPE
  Interventions: Device: MARPE (mini-screw assisted rapid palatal expansion)

INTERVENTIONS:
Device: MARPE (mini-screw assisted rapid palatal expansion) — MARPE (mini-screw assisted rapid palatal expansion) with two min screws in post-pubertal patients

SUMMARY:
a device is going to be placed in the palate to non-growing patients who are diagnosed to have a constricted maxillary arch and require an expansion of the maxillary arch in their treatment plan. the device is composed of two mini screws that will be placed in the palate which are connected to a hyrax with orthodontic bands on first maxillary molars. the activation of the device will be for 3 weeks 2 turns on the day of placement and 1 turn every day for 3 weeks. a CBCT x-ray will be taken before and after expansion to see the effect of MARPE on the mid-palatal suture.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of MARPE on MPS in post-pubertal patients using two mini-screws, evaluated by CBCT.

The sample will consist of 14 patients. They will be selected from the Orthodontic Department, Faculty of Dentistry, Mansuora University according to the following:

Inclusion criteria:

* Transverse maxillary deficiency with or without crossbite; who requires maxillary expansion in their treatment plan as described by Tamburino et al.19
* Age after 16.
* presence of first and second upper premolars and first upper molars
* No previous orthodontic treatment.
* Good oral hygiene and healthy periodontal tissue.
* No significant dentofacial anomalies, any bone defects, or systemic disease.
* Not being pregnant.
* All patients are signed a written consent after accepting the treatment plan.

Treatment procedure:

* First visit: Thorough explanation of procedures to the patient, clarifying all details and technical limitations and informing that failure may occur; placement of elastic separators on mesial and distal side of permanent maxillary first molars.
* Second visit: The elastic separators will be removed and a proper size of orthodontic bands will be placed in permanent maxillary first molars. After LA infiltration in the palate a two OrthoEasy Pal mini-screw from Forestadent size 8* 1.7 mm will be placed paramedian 3mm away from the midpalatal suture between the first and second premolar area,20 using a manual drive attachment for contra-angle handpiece and attached to OrthoEasy blade 10 mm Octagonal. After the placement of mini-screws in the desired location; two OrthoEasy Pal impression caps will be placed on the head of the mini-screws. After that, an impression will be taken using putty silicone impression material, the molar bands will be removed from patient's mouth using orthodontic band removal plier and placed in the impression tray. Also the impression cap will be removed from the patient's mouth and placed in the impression tray. Elastic separators on mesial and distal side of permanent maxillary first molars will be placed again.

The impression tray will be sent to the lab for MARPE fabrication.

Laboratory steps:

Before pouring the impression with regular white dental plaster, the impression caps will be removed from the impression tray and two OrthoEasy Pal lab analogs will be placed instead.

The impression will be poured with regular white dental plaster. 10 mm of palatal expansion screw from Forestadent will be selected according to the palatal width. The posterior wires will be bent to reach the orthodontic bands and soldered to it, while the anterior wires will be soldered to the OrthoEasy Pal abutment (flat profile) which will be placed on the cast on top of the duplicated mini-screw heads. followed by finishing and polishing of the device.

- Third visit: The elastic separators will be removed and the device will be placed to check its fitting. Once fitting is checked, cementation of the bands of the device to the first molar will be performed using glass ionomer cementation (GIC). After that, the OrthoEasy Pal abutments of the device will be retained to the mini-screws by OrthoEasy Pal Retaining screw using blade for OrthoEasy Pal retaining screw for contra-angle handpiece.

Immediate 2 turns activation will be made in the hyrax after fitting the appliance.

* The activation protocol of MARPE will be 1 turn per day for 3 weeks. After 3 weeks a cbct image will be taken to assess the MPS. Fixed appliance will be placed after 3-4 months period of retention.
* Activation will be discontinued when the lingual cusps of the upper first molars contacted the buccal cusps of the lower first molars.

Records:

For all patients the following records are made:

1. Photographs:

   1. Extraoral
   2. Intraoral
2. Upper and lower plaster casts.
3. Radiographs:

   1. Panoramic radiography.
   2. Lateral cephalometric.
   3. Cone-beam computed tomography systems (CBCT).

Photographs will be taken 3 times; pre-operative, after MARPE placement and after 3 weeks from the first activation

Upper and lower diagnostic casts will be taken once, pre- operative.

Lateral cephalometric and panoramic radiography will be taken once; pre operative. CBCT will be taken twice; pre-expansion and after 3 weeks from the first activation

1. Extra-oral and Intra-oral photographs:

   Extraoral photographs of the face in frontal and lateral views are taken. The frontal view is taken with the interpupillary line parallel to the floor and the midsagittal plane is perpendicular to the floor. The lateral view (left side) is taken after adjusting the Frankfort horizontal plane to be parallel to the the floor. on the other hand, the intraoral photographs are taken in frontal, lateral and occlusal views.
2. Upper and lower casts:

   Upper and lower impressions of the dental arches will be taken using Alginate impression material.They will be poured immediately in a white dental plaster. A wax bite is obtained in centric occlusion to orient the upper and lower casts. The models are identified with the name of the patient, date of birth, and date of taking the impression.
3. Radiographs:

   1. Lateral cephalometric radiograph: Lateral cephalometric radiographs are done before treatment as a diagnostic aids and to record the cervical vertebrae maturation.11
   2. Panoramic radiographs: Panoramic radiographs are taken before treatment as a diagnostic aids and to determine any pathological abnormalities that can hinder the study.
   3. Cone-beam computed tomography systems (CBCT): CBCT image (Soredex Cranex 3Dx) will be taken before expansion to record the stage of mid palatal suture21 and to assess the MPS. Another image will be taken after 3 weeks from the first activation for evaluating the mid-palatal suture.

At the following setting:

- Exposure time: 9 s, 4.0mA, 89kV, field of view [FOV]: 8*15 cm voxel size: 0.32 mm).

According to a previous puplished reseach, CBCT scans were taken before expansion (T1) and 1 week after active expansion (T2).22Another puplished research took CBCT scans before expansion (T1) and 10 days after active expansion (T2). 23 The CBCT setting will be reduced as much as possible with small field of view following the low dose protocol with the help of a radiologist from Mansuura university to ensure that the total radiation of repeated CBCT imaging during the experiment doesn't exceed the recommended annual dose limit (1 mSv).24

Digital Imaging and Communications in Medicine (DICOM) file image reconstruction and analysis will be performed with OsiriX Lite software.

CBCT analysis

For CBCT analysis; the following will be determined:

* dimensional reference planes for craniofacial structures orientation and to standardize linear measurements in the axial plane:

  - In the axial plane, the mid-palatine suture will be used.

  - In the mid-sagittal plane. the horizontal palatal plane will be the selected reference

  - In the coronal plane, the image was oriented perpendicular to the patient's midsagittal plane tangent to the most inferior level of nasal floor at the level of first molar where the crown and palatal root can be seen at their greatest length.
* After the image is oriented:

  1. For the pre-expansion images, the axial view will be chosen to determine the maturation stage of MPS and will be recorded.

  2. In both pre-expansion and after 3 weeks from the first activation images; points will be marked in the axial plane at 3 different locations assisted from coronal plane: first premolar, second premolar and first molar.
* For the first premolar and the first molar: points will be made at the most anterior section where the crown and palatal root can be seen at their greatest length.

For the second premolar: in the most anterior section showing maximum length of its root.

• Measuring the distance between the external right and left maxilla edges in the axial view before expansion and after 3 weeks from the first activation

ELIGIBILITY:
Inclusion Criteria:

* Transverse maxillary deficiency with or without crossbite; who requires maxillary expansion in their treatment plan as described by Tamburino et al.3
* Age after 16.
* Presence of first and second upper premolars and first upper molars.
* No previous orthodontic treatment.
* Good oral hygiene and healthy periodontal tissue.
* No significant dentofacial anomalies, any bone defects, or systemic disease.
* Not being pregnant.
* All patients were signed a written consent after accepting the treatment plan.

Exclusion Criteria

* Patients under the age of 16 years.
* Absence of first and second upper premolars and first upper molars.
* Previous orthodontic treatment
* Periodontal disease and poor oral hygiene
* significant dentofacial anomalies, any bone defects, or systemic disease.
* Pregnant
* Those who did not consent to participate in this study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
CBCT analysis : the mid palatal suture opening will be assessed from the axial slice. | 3 weeks in each participant
  CBCT analysis: the mid palatal suture opening will be measures in millimetres at three different sites ( first premolar , second premolar, first molar). the metric measure will be placed at the two ends of the mid palatal suture

CONTACTS AND LOCATIONS:
Locations (1):
- Mansura University, Faculty of Dentistry, Al Mansurah, Al Dakhelia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT07075211/Prot_SAP_000.pdf